CLINICAL TRIAL: NCT04501107
Title: A Randomised, Double Blind, Crossover Euglycaemic Clamp Trial to Compare BioChaperone Insulin Lispro Formulations With US Approved Humalog® and With EU Approved Humalog® in Patients With Type 1 Diabetes Mellitus
Brief Title: A Trial to Compare BioChaperone Insulin Lispro Formulations With US Approved Humalog® and With EU Approved Humalog® in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT037-ADO02
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; signal peptide peptidase; IGF2BP2 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BioChaperone insulin lispro reconstituted with Humalog® (IMP1) (Experimental): Subcutaneous administration of Biochaperone insulin lispro formulation made from a freeze-dried of BioChaperone reconstituted with Humalog® at a dose of 0.2 U/Kg Body Weight (BW).
  Interventions: Drug: Administration of BioChaperone insulin lispro reconstituted with Humalog® (IMP1)
- Ready-to-use BioChaperone insulin lispro (IMP2) (Experimental): Subcutaneous administration of ready-to-use Biochaperone insulin lispro formulation at a dose of 0.2 U/Kg BW.
  Interventions: Drug: Administration of Ready-to-use BioChaperone insulin lispro (IMP2)
- US-approved Humalog® (IMP3) (Active Comparator): Subcutaneous administration of US-approved Humalog® at a dose of 0.2 U/Kg BW.
  Interventions: Drug: Administration of US-approved Humalog® (IMP3)
- EU-approved Humalog® (IMP4) (Active Comparator): Subcutaneous administration of EU-approved Humalog® at a dose of 0.2 U/Kg BW.
  Interventions: Drug: Administration of EU-approved Humalog® (IMP4)

INTERVENTIONS:
Drug: Administration of BioChaperone insulin lispro reconstituted with Humalog® (IMP1) — Administration of IMP1 during a 12-hour euglycaemic clamp.
  Arms: BioChaperone insulin lispro reconstituted with Humalog® (IMP1)
Drug: Administration of Ready-to-use BioChaperone insulin lispro (IMP2) — Administration of IMP2 during a 12-hour euglycaemic clamp.
  Arms: Ready-to-use BioChaperone insulin lispro (IMP2)
Drug: Administration of US-approved Humalog® (IMP3) — Administration of IMP3 during a 12-hour euglycaemic clamp.
  Arms: US-approved Humalog® (IMP3)
Drug: Administration of EU-approved Humalog® (IMP4) — Administration of IMP4 during a 12-hour euglycaemic clamp.
  Arms: EU-approved Humalog® (IMP4)

SUMMARY:
This is a single-centre, randomised, double-blind, 4-way crossover, 4-treatment, euglycaemic clamp study in subjects with Type 1 Diabetes Mellitus (T1DM). Each subject will be randomly allocated to one of four treatment sequences. Each sequence comprises one single dose of each of four IMPs. IMP1 and IMP2 are BioChaperone lispro formulations. They have the same composition and correspond to different development stages of a unique product which is BioChaperone insulin lispro; between them, improvements were made to prepare industrial production. Comparators (IMP3 and IMP4) are US-approved Humalog® and EU-approved Humalog®. All IMPs will be dosed at 0.2 U/Kg of insulin lispro on 4 dosing visits separated by a washout period of 5 to 15 days.

The trial will compare the characteristics of BioChaperone insulin lispro fully liquid (IMP2) formulation to US-approved Humalog and EU-approved Humalog.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 Diabetes Mellitus
* Body Mass Index (BMI) between 18.5 and 28.5 kg/m^2, both inclusive
* HbA1c <= 75 mmol/mol (<=9.0%).
* Fasting negative C-peptide (<= 0.30 nmol/L).
* Total insulin dose of < 1.2 (I)U/kg/day.
* Stable insulin regimen (with respect to safety of the subject and scientific integrity of the study) using continuous subcutaneous insulin infusion (CSII) or multiple daily insulin injections (MDI) for at least 2 months.

Exclusion Criteria:

* Known or suspected hypersensitivity to IMP(s) or related products.
* Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomisation in this trial.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator.
* Any history or presence of clinically relevant comorbidity capable of constituting a risk for the subject when participating in the trial or of interfering with the interpretation of data.
* Signs of acute illness as judged by the Investigator.
* Any serious systemic infectious disease during four weeks prior to first dosing of the trial drug, as judged by the Investigator.
* Clinically significant abnormal screening laboratory tests, as judged by the Investigator.
* Proliferative retinopathy or maculopathy as judged by the Investigator based on a recent (<1.5 years) ophthalmologic examination.
* Use of oral antidiabetic drugs (OADs) and/or GLP-1 receptor agonists within 3 months prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
AUCGIR.0-12h | From t=0 to t=12 hours after IMP administration
  Area under the glucose infusion rate-time curve from time 0 until end of clamp
AUCGIR.0-1h | From t=0 to t=1 hour after IMP administration
  Area under the glucose infusion rate-time curve from time 0 to 1 hour after IMP administration
AUCLIS.0-12h | From t=0 to t=12 hours after IMP administration
  Area under the insulin lispro concentration-time curve from 0 hours to 12 hours after dose administration
AUCLIS.0-1h | From t=0 to t=1 hour after IMP administration
  Area under the insulin lispro concentration-time curve from 0 hours to 1 hour after dose administration

SECONDARY OUTCOMES:
tmax.LIS | From t=0 to t=12 hours after IMP administration
  Time to maximum observed insulin lispro concentration
Cmax.LIS | From t=0 to t=12 hours after IMP administration
  Maximum observed insulin lispro concentration
AUCLIS.2-6h | From t=2 to t=6hours after IMP administration
  Area under the insulin lispro concentration-time curve from 2 hour to 6 hour after dose administration
t50%-LIS (early) | From t=0 to t=12 hours after IMP administration
  Time to half-maximum before Cmax.LIS
tmax.GIR | From t=0 to t=12 hours after IMP administration
  Time to maximum glucose infusion rate
GIRmax | From t=0 to t=12 hours after IMP administration
  Maximum glucose infusion rate
AUCGIR.4-8h | From t=4 to t=8 hours after IMP administration
  Area under the glucose infusion rate-time curve from 4 to 8 hours after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Baumgaertner, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Mainz, Germany